CLINICAL TRIAL: NCT00942773
Title: Clinical Trials to Evaluate the Influence of CYP2C19 Genotype and Drug-drug Interactions on the Pharmacokinetics of Voriconazole in Healthy Korean Male Volunteers (Part A)
Brief Title: Influence of CYP2C19 Genotype on the Pharmacokinetics (PK) of Voriconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: In-Jin Jang, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SNUCPT09_Vori2C19_A
Record Dates: First submitted 2009-07-14; First posted 2009-07-21 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Healthy volunteer
MeSH Terms: interventions — Voriconazole

ARMS (3):
- CYP2C19 extensive metabolizer (Active Comparator)
  Interventions: Drug: Voriconazole
- CYP2C19 heterozygous extensive metabolizer (Active Comparator)
  Interventions: Drug: Voriconazole
- CYP2C19 poor metabolizer (Active Comparator)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
The purpose of this study is to:

* Evaluate the influence of CYP2C19 genotype on PK profiles of voriconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 20 - 50 years.
2. A body mass index (BMI) in the range 17-28 kg/m2.
3. Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully. informed about the study procedures.

Exclusion Criteria:

1. Presence or history of severe adverse reaction to any drug or a history of severe allergic disease.
2. Clinically relevant abnormal medical history that could interfere with the objectives of the study.
3. Presence or history of eye disease or eye field defect.
4. A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug.
5. A subject whose liver function test (AST, ALT, GGT, ALP, LDH) result is over 1.25 times of upper limit of normal range.
6. A subject whose SBP is over 140 mmHg or below 90 mmHg and DBP is over 100 mmHg or below 50 mmHg.
7. Presence or history of drug abuse.
8. Participation in other clinical trial within 2 months.
9. Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication within 1 week before first dose.
10. Blood donation during 2 months or apheresis during 1 month before the study.
11. Presence or history of alcohol abuse.
12. Smoking of more than 10 cigarettes/day.
13. Use of grapefruit juice, xanthine containing beverage, alcohol or smoking during restriction period.
14. Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of voriconazole

SECONDARY OUTCOMES:
Adverse events collected by investigator questionnaire and subjects spontaneous report
12-lead ECG
Clinical laboratory test
Vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee S, Gu N, Kim BH, Lim KS, Shin SG, Jang IJ, Yu KS. Pharmacokinetic and pharmacodynamic properties of the calcimimetic agent cinacalcet (KRN1493) in healthy male Korean subjects: a randomized, open-label, single ascending-dose, parallel-group study. Clin Ther. 2012 May;34(5):1160-9. doi: 10.1016/j.clinthera.2012.03.058. Epub 2012 Apr 13. PMID 22503212
- [Derived] Lee S, Kim BH, Nam WS, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Effect of CYP2C19 polymorphism on the pharmacokinetics of voriconazole after single and multiple doses in healthy volunteers. J Clin Pharmacol. 2012 Feb;52(2):195-203. doi: 10.1177/0091270010395510. PMID 21383338